CLINICAL TRIAL: NCT03685344
Title: A Phase 1 Open-Label Study to Evaluate the Safety and Antitumor Activity of Loncastuximab Tesirine and Durvalumab in Patients With Advanced Diffuse Large B-Cell Lymphoma, Mantle Cell Lymphoma, or Follicular Lymphoma
Brief Title: Safety and Antitumor Activity Study of Loncastuximab Tesirine and Durvalumab in Diffuse Large B-Cell, Mantle Cell, or Follicular Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: In a limited number of patients, no additional activity was evident for the combination vs. loncastuximab tesirine monotherapy.
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-104; 2018-002670-43 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-09-26 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma
Keywords: Loncastuximab Tesirine in Combination with Durvalumab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular | interventions — loncastuximab tesirine; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCT-402 (Experimental): Dose escalation phase: Ascending doses of Loncastuximab tesirine will be administered using a traditional 3+3 design. Dose level 1: 90 µg/kg, every 3 weeks (Q3W). Dose level 2: 120 µg/kg, Q3W. Dose level 3: 150 µg/kg, Q3W. Loncastuximab tesirine will be given for 2 doses, 3 weeks apart.
  Dose expansion phase: Loncastuximab tesirine will be administered at the recommended dose determined in the dose escalation phase. Durvalumab will also be administered at a dose of 1500 mg once every 4 weeks (Q4W) throughout the dose escalation phase and dose expansion phase.
  Interventions: Drug: Loncastuximab Tesirine and Durvalumab

INTERVENTIONS:
Drug: Loncastuximab Tesirine and Durvalumab — intravenous infusion
  Other Names: ADCT-402 in combination with Durvalumab; Zynlonta

SUMMARY:
The purpose of this phase 1 study is to evaluate the safety and anti-tumor activity of Loncastuximab Tesirine (ADCT-402) and Durvalumab in participants with Advanced Diffuse Large B-Cell Lymphoma, Mantle Cell Lymphoma, or Follicular Lymphoma

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, single-arm combination study with a dose escalation phase (Part 1) followed by a dose expansion phase (Part 2). The study will enroll approximately 75 participants.

A standard 3+3 dose escalation design will be used for Part 1. The DLT period will be the 21 days after the first durvalumab dose.

Part 2 will consist of up to 3 expansion cohorts, one for DLBCL, one for MCL, and one for FL. Each cohort will be approximately 20 participants treated at the dose determined in Part 1.

The study will include a Screening Period (of up to 28 days), a Treatment Period (cycles of 3, 6, and 4 weeks), and a Follow-up Period (approximately every 12 week visits for up to 2 years after treatment discontinuation).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older
2. Pathologic diagnosis of DLBCL, MCL, or FL
3. Participants must have relapsed or refractory disease and have failed or been intolerant to standard therapy
4. Participants who have received previous CD19-directed therapy must have a biopsy that shows CD19 expression after completion of the CD19-directed therapy
5. Measurable disease as defined by the 2014 Lugano Classification
6. Participants must be willing to undergo tumor biopsy
7. ECOG performance status 0-1
8. Screening laboratory values within the following parameters:

   1. Absolute neutrophil count (ANC) ≥1.0 × 103/µL (off growth factors at least 72 hours)
   2. Platelet count ≥75 × 103/µL without transfusion in the past 7 days
   3. Hemoglobin ≥9.0 g/dL (5.59 mmol/L), transfusion allowed
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and GGT ≤2.5 × the upper limit of normal (ULN)
   5. Total bilirubin ≤1.5 × ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 × ULN)
   6. Blood creatinine ≤1.5 × ULN or calculated creatinine clearance ≥60 mL/min by the Cockcroft-Gault equation
9. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test within 3 days prior to start of study drug on C1D1 for women of childbearing potential
10. Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the last dose of study therapy. Men with female partners who are of childbearing potential must agree that they will use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the patient receives his last dose of study therapy

Exclusion Criteria:

1. Known history of hypersensitivity to or positive serum human ADA to a CD19 antibody.
2. Previous therapy with any checkpoint inhibitor
3. Autologous stem cell transplant within 100 days prior to start of study drug (C1D1)
4. History of allogenic stem cell transplant
5. History of solid organ transplant
6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   1. Participants with vitiligo or alopecia
   2. Participants with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Participants without active disease in the last 5 years may be included but only after consultation with the Study Physician
   5. Participants with celiac disease controlled by diet alone
7. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice)
8. Known seropositive and requiring anti-viral therapy for human immunodeficiency (HIV) virus, hepatitis B virus (HBV), or hepatitis C virus (HCV)
9. History of Stevens-Johnson syndrome or toxic epidermal necrolysis
10. Lymphoma with active central nervous system (CNS) involvement at the time of screening, including leptomeningeal disease
11. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
12. Breastfeeding or pregnant
13. Significant medical comorbidities, including but not limited to, uncontrolled hypertension (blood pressure [BP] ≥160/100 mmHg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes, or severe chronic pulmonary disease
14. Radiotherapy, chemotherapy, or other anti-neoplastic therapy within 14 days prior to start of study drug (C1D1), except shorter if approved by the Sponsor.
15. Major surgery within 28 days prior to start of study drug (C1D1), except shorter if approved by the Sponsor. Note: Local surgery of isolated lesions for palliative intent is acceptable.
16. Use of any other experimental medication within 14 days prior to start of study drug (C1D1)
17. Planned live vaccine administration after starting study drug (C1D1)
18. Failure to recover to Grade ≤1 (Common Terminology Criteria for Adverse Events [CTCAE] version 4.0) from acute non-hematologic toxicity (Grade ≤2 neuropathy or alopecia) due to previous therapy prior to screening.
19. Congenital long QT syndrome or a corrected QTcF interval of >470 ms at screening (unless secondary to pacemaker or bundle branch block)
20. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of investigational product and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease 21. History of active primary immunodeficiency
21. History of active primary immunodeficiency or any other significant medical illness, abnormality, or condition that would, in the Investigator's judgement, make the patient inappropriate for study participation or put the participant at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCH-MHS Memorial Hospital Centeral, Colorado Springs, Colorado
  - University of Florida Health Shands Cancer Hospital, Gainesville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Icahm School of Medicine at Mount Sinai, New York, New York
  - Baylor University Medical Center, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon Pabellón de Oncología, Madrid
  - Hospital Universitario Fundación Jiménez Díaz Unidad de Limfomas Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen Macarena Servicio Oncologia Medica, Seville
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 participants were enrolled at 5 sites in the United States and 3 sites in Spain between February 2019 and October 2020.
Pre-assignment Details: 16 participants had signed informed consent, however 3 were considered screen failures. The remaining 13 participants were enrolled and received study treatment.
Groups:
- Dose Escalation: Loncastuximab Tesirine 90 μg/kg: Participants received loncastuximab tesirine as an intravenous (IV) infusion at a dose of 90 micrograms per kilogram (μg/kg) every 3 weeks (Q3W) on Day 1 of Cycles 1 and 2. Cycle 1 was 3 weeks long and Cycle 2 was 6 weeks long. Participants with a partial response (PR) or stable disease (SD) at Week 15 received an additional 2 doses of loncastuximab tesirine on Day 8 of Cycles 5 and 6. All cycles other than Cycles 1 and 2 were 4 weeks long. Participants also received durvalumab as an IV infusion at a dose of 1500 milligrams (mg) on Day 8 of Cycle 1 and Day 15 of Cycle 2, then on Day 1 of subsequent cycles.
- Dose Escalation: Loncastuximab Tesirine 120 μg/kg: Participants received loncastuximab tesirine as an IV infusion at a dose of 120 μg/kg Q3W on Day 1 of Cycles 1 and 2. Cycle 1 was 3 weeks long and Cycle 2 was 6 weeks long. Participants with a PR or SD at Week 15 received an additional 2 doses of loncastuximab tesirine on Day 8 of Cycles 5 and 6. All cycles other than Cycles 1 and 2 were 4 weeks long. Participants also received durvalumab as an IV infusion at a dose of 1500 mg on Day 8 of Cycle 1 and Day 15 of Cycle 2, then on Day 1 of subsequent cycles.
- Dose Escalation: Loncastuximab Tesirine 150 μg/kg: Participants received loncastuximab tesirine as an IV infusion at a dose of 150 μg/kg Q3W on Day 1 of Cycles 1 and 2. Cycle 1 was 3 weeks long and Cycle 2 was 6 weeks long. Participants with a PR or SD at Week 15 received an additional 2 doses of loncastuximab tesirine on Day 8 of Cycles 5 and 6. All cycles other than Cycles 1 and 2 were 4 weeks long. Participants also received durvalumab as an IV infusion at a dose of 1500 mg on Day 8 of Cycle 1 and Day 15 of Cycle 2, then on Day 1 of subsequent cycles.
- Dose Expansion: Loncastuximab Tesirine: The dose expansion phase was planned to consist of participants with diffuse large B-cell lymphoma, participants with mantle cell lymphoma and participants with follicular lymphoma.
  Participants were planned to receive loncastuximab tesirine as an IV infusion at the maximum tolerated dose (MTD) determined in the dose escalation part and durvalumab as an IV infusion at a dose of 1500 mg on Day 8 of Cycle 1 and Day 15 of Cycle 2, then on Day 1 of subsequent cycles.
  The study was terminated during the dose escalation part of the study and the dose expansion part was not initiated.
Period: Overall Study
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Started | 3 | 3 | 7 | 0
Received Treatment | 3 | 3 | 7 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 7 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 5 | 0
Not completed — Death | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set - All participants who received the study drug. The study was terminated during the dose escalation part of the study and the dose expansion part was not initiated, therefore data is only available for the dose escalation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine | Total
Number analyzed (Participants) | 3 | 3 | 7 | 0 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (15.00) | 74.0 (2.00) | 63.0 (16.94) |  | 66.2 (14.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 |  | 6
  Male | 2 | 0 | 5 |  | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 |  | 4
  Not Hispanic or Latino | 1 | 3 | 5 |  | 9
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 0 |  | 0
  White | 3 | 3 | 5 |  | 11
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an adverse event (AE) that occurred or worsened in the period extending from the first dose of study drugs to 30 days after the last dose of study drugs or initiation of new anti-cancer therapy (whichever occurred earlier).
  Evaluation of TEAEs included the number of participants with at least one: TEAE, serious TEAE and grade ≥3 TEAE as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
  CTCAE grading scale:
  * Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living.
  * Grade 4 = Life-threatening consequences; urgent intervention indicated.
  * Grade 5 = Death related to AE.
  Clinically significant changes from baseline for safety laboratory values, vital sign measurements and electrocardiograms (ECGs) were recorded as TEAEs.
Time Frame: Day 1 to 30 days after the last dose of study drugs (maximum treatment duration at study termination was 336 days)
Population: Safety analysis set - All participants who received the study drug. The study was terminated prior to initiation of the dose expansion, so results are only presented for the dose escalation.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
Participants
  TEAE | 3 | 3 | 7 |
  Serious TEAE | 1 | 2 | 1 |
  CTCAE Grade ≥3 TEAE | 2 | 2 | 5 |

2. Primary Outcome: Number of Participants With a Dose-limiting Toxicity
Description: DLTs were defined as specific events which occurred in the 21-day DLT evaluation period of the dose escalation part, except any events that were clearly due to underlying disease or extraneous causes. The grading and severity of events were based on the guidelines provided in the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 21 days after first dose of durvalumab (Day 8 to Day 29)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
Participants | 0 | 0 | 0 |

3. Primary Outcome: Number of Participants With a Treatment-emergent Adverse Event Leading to Dose Interruption or Reduction
Time Frame: Day 1 to end of treatment (maximum treatment duration at study termination was 336 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
Participants
  Loncastuximab Tesirine: Dose Interruption | 0 | 0 | 0 |
  Loncastuximab Tesirine: Dose Reduction | 0 | 0 | 0 |
  Durvalumab: Dose Interruption | 0 | 0 | 0 |
  Durvalumab: Dose Reduction | 0 | 0 | 0 |

4. Primary Outcome: Number of Participants With Changes From Baseline on the Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Eastern Cooperative Oncology Group (ECOG) performance status was scored on a 6-point scale where higher scores indicate a worse outcome. ECOG scores included the following:
  * 0 = fully active, able to carry on all pre-disease performance without restriction
  * 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * 2 = ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  * 3 = capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  * 4 = completely disabled; cannot carry on any self-care; totally confined to bed or chair
  * 5 = dead
Time Frame: Day 1 to end of treatment (maximum treatment duration at study termination was 336 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
Participants | 2 | 0 | 1 |

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR according to the 2014 Lugano classification as determined by the investigator. Overall response rate was the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR).
  CR was defined as achieving each of the following:
  * Complete metabolic response.
  * Complete radiologic response (target node regress to <1.5 cm, no non-measured lesions, no organ enlargement, no new lesions and normal bone marrow morphology).
  PR was defined as achieving each of the following:
  * Partial metabolic response (findings indicate residual disease).
  * Partial remission (>50% decrease in target measurable nodes, regression/ absence/ no increase of non-measured lesions, spleen regressed by >50% in length and no new lesions).
Time Frame: Up to 1.5 years
Population: Efficacy analysis set - All participants who received at least one dose of study drug, had valid baseline disease assessment(s) and at least one valid post-baseline disease assessment. Participants who did not have a post-baseline assessment due to early clinical progression or death (after receiving study drug) were also included. The study was terminated prior to initiation of the dose expansion, so results are only presented for the dose escalation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 2 | 7 | 0
percentage of participants | 33.3 [0.8 to 90.6] | 100 [15.8 to 100] | 71.4 [29.0 to 96.3] |

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the documentation of first tumor response (CR or PR) to disease progression or death.
  CR was defined as achieving each of the following:
  * Complete metabolic response.
  * Complete radiologic response (target node regress to <1.5 cm, no non-measured lesions, no organ enlargement, no new lesions and normal bone marrow morphology).
  PR was defined as achieving each of the following:
  * Partial metabolic response (findings indicate residual disease).
  * Partial remission (>50% decrease in target measurable nodes, regression/ absence/ no increase of non-measured lesions, spleen regressed by >50% in length and no new lesions).
Time Frame: Up to 1.5 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
months | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. |

7. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR was defined as the percentage of participants with a BOR of CR, according to the 2014 Lugano classification, as determined by the investigator.
  CR was defined as achieving each of the following:
  * Complete metabolic response.
  * Complete radiologic response (target node regress to <1.5 cm, no non-measured lesions, no organ enlargement, no new lesions and normal bone marrow morphology).
Time Frame: Up to 1.5 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 2 | 7 | 0
percentage of participants | 0 [NA to NA] — 0 participants had a BOR of CR. | 50 [1.3 to 98.7] | 0 [NA to NA] — 0 participants had a BOR of CR. |

8. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined as the time from the documentation of CR to disease progression or death.
  CR was defined as achieving each of the following:
  * Complete metabolic response.
  * Complete radiologic response (target node regress to <1.5 cm, no non-measured lesions, no organ enlargement, no new lesions and normal bone marrow morphology).
  Disease progression was defined as progressive metabolic disease and one of the following:
  * Target node progression.
  * An individual extranodal lesion must be abnormal with length > 1.5cm and/or increase of length > 50%.
  * New or clear progression of non-measured lesions.
  * Regrowth of previously resolved lesions or new nodes >1.5 cm in length.
  * New or recurrent bone marrow involvement.
Time Frame: Up to 1.5 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 2 | 7 | 0
months | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. |

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time between start of treatment and the first documentation of progression, or death.
  Disease progression was defined as progressive metabolic disease and one of the following:
  * Target node progression.
  * An individual extranodal lesion must be abnormal with length > 1.5cm and/or increase of length > 50%.
  * New or clear progression of non-measured lesions.
  * Regrowth of previously resolved lesions or new nodes >1.5 cm in length.
  * New or recurrent bone marrow involvement.
Time Frame: Up to 1.5 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 2 | 7 | 0
months | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. |

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the start of treatment and death from any cause.
Time Frame: Up to 1.5 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 2 | 7 | 0
months | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. | NA (NA) — Due to early termination, there was an insufficient number of participants to be able to analyze this endpoint. |

11. Secondary Outcome: Maximum Concentration (Cmax) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Description: Cmax of loncastuximab tesirine conjugated antibody and total antibody was calculated for Cycles 1 and 2. Cmax of warhead SG3199 was only calculated for Cycle 1 as data was not collected for Cycle 2.
Time Frame: Cycles 1 and 2 (where Cycle 1 was 4 weeks long and Cycle 2 was 6 weeks long): Day 1 pre-dose and at 0.5 and 4 hours post-dose, Day 8 and Day 15
Population: Pharmacokinetics (PK) population - All participants with at least one pre- Cycle 1 Day 1 (C1D1) and one post-dose valid assessment. The study was terminated prior to initiation of the dose expansion, so results are only presented for the dose escalation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
nanograms per milliliter (ng/mL)
  Cycle 1 - Conjugated Antibody | 540 (52.4) | 1683 (22.6) | 1980 (30.6) |
  Cycle 1 - Total Antibody | 1001 (51.6) | 3122 (16.7) | 2966 (25.4) |
  Cycle 1 - SG3199: number analyzed (Participants) | 0 | 0 | 3 | 0
  Cycle 1 - SG3199 |  |  | 0.0350 (58.5) |
  Cycle 2 - Conjugated Antibody: number analyzed (Participants) | 3 | 3 | 5 | 0
  Cycle 2 - Conjugated Antibody | 621 (48.7) | 1946 (33.5) | 1582 (31.7) |
  Cycle 2 - Total Antibody: number analyzed (Participants) | 3 | 3 | 5 | 0
  Cycle 2 - Total Antibody | 1228 (44.6) | 3510 (23.9) | 2899 (29.3) |

12. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Description: AUC0-last of loncastuximab tesirine conjugated antibody and total antibody was calculated for Cycles 1 and 2. AUC0-last of warhead SG3199 was only calculated for Cycle 1 as data was not collected for Cycle 2.
Time Frame: as for outcome 11
Population: PK population - All participants with at least one pre- C1D1 and one post-dose valid assessment. The study was terminated prior to initiation of the dose expansion, so results are only presented for the dose escalation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram days per milliliter (day*ng/mL)
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
nanogram days per milliliter (day*ng/mL)
  Cycle 1 - Conjugated Antibody | 4265 (52.5) | 17217 (32.7) | 5763 (253) |
  Cycle 1 - Total Antibody | 7603 (35.0) | 29456 (34.3) | 3682 (917) |
  Cycle 1 - SG3199: number analyzed (Participants) | 0 | 0 | 3 | 0
  Cycle 1 - SG3199 |  |  | 0.00300 (61.9) |
  Cycle 2 - Conjugated Antibody: number analyzed (Participants) | 3 | 3 | 5 | 0
  Cycle 2 - Conjugated Antibody | 5305 (24.9) | 5390 (1410) | 7588 (61.7) |
  Cycle 2 - Total Antibody: number analyzed (Participants) | 3 | 3 | 5 | 0
  Cycle 2 - Total Antibody | 10388 (21.1) | 9122 (1485) | 13264 (67.9) |

13. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Description: AUCinf of loncastuximab tesirine conjugated antibody and total antibody was calculated for Cycles 1 and 2. AUCinf of warhead SG3199 was only calculated for Cycle 1 as data was not collected for Cycle 2.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram days per milliliter (day*ng/mL)
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 2 | 2 | 2 | 0
nanogram days per milliliter (day*ng/mL)
  Cycle 1 - Conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 1 - Total Antibody: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 1 - Total Antibody |  |  | 15954 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. |
  Cycle 1 - SG3199: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 2 - Conjugated Antibody | 5461 (64.5) | 18182 (15.3) | 8504 (41.4) |
  Cycle 2 - Total Antibody: number analyzed (Participants) | 1 | 1 | 2 | 0
  Cycle 2 - Total Antibody | 7710 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 27875 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 15382 (54.0) |

14. Secondary Outcome: Apparent Terminal Half-life (Thalf) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Description: Thalf of loncastuximab tesirine conjugated antibody and total antibody was calculated for Cycles 1 and 2. Thalf of warhead SG3199 was only calculated for Cycle 1 as data was not collected for Cycle 2.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 2 | 2 | 2 | 0
day
  Cycle 1 - Conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 1 - Total Antibody: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 1 - Total Antibody |  |  | 8.13 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. |
  Cycle 1 - SG3199: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 2 - Conjugated Antibody | 8.84 (33.6) | 16.9 (54.9) | 5.93 (213) |
  Cycle 2 - Total Antibody: number analyzed (Participants) | 1 | 1 | 2 | 0
  Cycle 2 - Total Antibody | 15.1 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 33.9 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 6.28 (180) |

15. Secondary Outcome: Apparent Clearance (CL) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Description: CL for Cycle 2 reflects steady-state clearance. CL of loncastuximab tesirine conjugated antibody and total antibody was calculated for Cycles 1 and 2.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per day (L/day)
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 2 | 2 | 2 | 0
liters per day (L/day)
  Cycle 1 - Conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 1 - Total Antibody: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 1 - Total Antibody |  |  | 0.846 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. |
  Cycle 1 - SG3199: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 2 - Conjugated Antibody | 0.927 (50.7) | 0.319 (6.31) | 1.33 (36.4) |
  Cycle 2 - Total Antibody: number analyzed (Participants) | 1 | 1 | 2 | 0
  Cycle 2 - Total Antibody | 0.720 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 0.212 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 0.872 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. |

16. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Description: Vss of loncastuximab tesirine conjugated antibody and total antibody was calculated for Cycles 1 and 2.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 2 | 2 | 2 | 0
liters (L)
  Cycle 1 - Conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 1 - Total Antibody: number analyzed (Participants) | 0 | 0 | 1 | 0
  Cycle 1 - Total Antibody |  |  | 9.39 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. |
  Cycle 1 - SG3199: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 2 - Conjugated Antibody | 11.3 (94.4) | 7.36 (38.7) | 6.95 (270) |
  Cycle 2 - Total Antibody: number analyzed (Participants) | 1 | 1 | 2 | 0
  Cycle 2 - Total Antibody | 13.7 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 8.61 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 5.14 (171) |

17. Secondary Outcome: Accumulation Index (AI) of Loncastuximab Tesirine Conjugated Antibody and Total Antibody
Description: AI is the ratio of drug accumulation after repeated administration compared to a single dose. AI of loncastuximab tesirine conjugated antibody and total antibody was calculated from Cycles 1 and 2.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 2 | 2 | 2 | 0
ratio
  Cycle 1 - Conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 1 - Total Antibody: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cycle 2 - Conjugated Antibody | 1.25 (12.9) | 1.77 (33.0) | 1.27 (34.4) |
  Cycle 2 - Total Antibody: number analyzed (Participants) | 1 | 1 | 2 | 0
  Cycle 2 - Total Antibody | 1.62 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 2.87 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 1.26 (33.3) |

18. Secondary Outcome: Number of Participants With an Anti-drug Antibody (ADA) Response to Loncastuximab Tesirine
Description: Detection of ADAs were performed by using a screening assay for identification of antibody positive samples/patients, a confirmation assay, and titer assessment, and were performed using the Meso-Scale Discovery Electrochemiluminescence platform.
Time Frame: Cycle 1 (= 3 weeks): Day 1 pre-dose & Day 15; Cycles 2, 3, 5, 6, & 7 (Cycle 2 = 6 weeks, other cycles = 4 weeks): Day 1 pre-dose; 30 days after last dose of study drugs
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
Number analyzed (Participants) | 3 | 3 | 7 | 0
Participants | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: Day 1 up to end of follow-up (maximum duration was 1.5 years)
Description: TEAEs collected up to 30 days after last dose of study drug or initiation of new anti-cancer therapy. The only AEs collected beyond that were treatment related SAEs and ACM for up to 1.5 years
Arm/Group | Dose Escalation: Loncastuximab Tesirine 90 μg/kg | Dose Escalation: Loncastuximab Tesirine 120 μg/kg | Dose Escalation: Loncastuximab Tesirine 150 μg/kg | Dose Expansion: Loncastuximab Tesirine
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/7 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Loncastuximab Tesirine 90 μg/kg (N=3) | Dose Escalation: Loncastuximab Tesirine 120 μg/kg (N=3) | Dose Escalation: Loncastuximab Tesirine 150 μg/kg (N=7) | Dose Expansion: Loncastuximab Tesirine (N=0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Loncastuximab Tesirine 90 μg/kg (N=3) | Dose Escalation: Loncastuximab Tesirine 120 μg/kg (N=3) | Dose Escalation: Loncastuximab Tesirine 150 μg/kg (N=7) | Dose Expansion: Loncastuximab Tesirine (N=0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (10) | 1 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03685344/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03685344/SAP_001.pdf